CLINICAL TRIAL: NCT00387569
Title: A Randomized, Observer-Blinded, Parallel-Group, Active-Control, Phase 1/2 Trial of the Safety, Immunogenicity, and Tolerability of 20 µg, 60 µg, and 200 µg of Meningococcal Group B rLP2086 Vaccine in Healthy Adolescents Aged 10 to 12 Years
Brief Title: Study Evaluating Safety & Immunogenicity of rLP2086 Vaccine in Healthy Toddlers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 6108A1-502
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-05

CONDITIONS: Healthy
Keywords: Toddlers; Vaccine; Safety

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Experimental (20ug); Active Comparator/Placebo
  Interventions: Biological: MnB vaccine rLP8026
- Cohort 2 (Experimental): Experimental (60ug); Active Comparator/Placebo
  Interventions: Biological: MnB vaccine rLP8026
- Cohort 3 (Experimental): Experimental (200ug); Active Comparator/Placebo
  Interventions: Biological: MnB vaccine rLP8026

INTERVENTIONS:
Biological: MnB vaccine rLP8026 — MnB vaccine at 20ug dose (0,1,6 months) or control (Hepatitis A vaccine, placebo, Hepatitis A vaccine at 0,1,6 months, respectively)
  Arms: Cohort 1
Biological: MnB vaccine rLP8026 — MnB vaccine at 60ug dose (0,1,6 months) or control (Hepatitis A vaccine, placebo, Hepatitis A vaccine at 0,1,6 months, respectively)
  Arms: Cohort 2
Biological: MnB vaccine rLP8026 — MnB vaccine at 200ug dose (0,1,6 months) or control (Hepatitis A vaccine, placebo, Hepatitis A vaccine at 0,1,6 months, respectively)
  Arms: Cohort 3

SUMMARY:
A study to assess the safety of an investigational meningitis vaccine in toddlers and their immune response to it.

ELIGIBILITY:
Inclusion Criteria

* Aged 18- to 36-months
* Healthy male or female subjects

Exclusion Criteria

* Prior vaccination with a serogroup B meningococcal vaccine
* Prior history of any invasive meningococcal disease

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 99 (Estimated)
Dates: Start 2006-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Local and systemic reactions through 14 days post-injection; Vaccinations at 0,1,6 months | Vaccinations at 0,1,6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Australia, medinfo@wyeth.com
Locations (1):
- Perth, Western Australia, Australia